CLINICAL TRIAL: NCT02160119
Title: Emotional and Change-related Attention in Autism
Acronym: AUTATTEN
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C13-26; 2013-A01315-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-06-03; First posted 2014-06-10 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2021-08

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorders; Emotion; Attention; Event-related potential; Functional neuroimaging; Diffusion Tensor Imaging; Development
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Diffusion Tensor Imaging; Evoked Potentials

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Controls
  Interventions: Other: MRI-based techniques; Other: EEG
- Autism Spectrum Disorders
  Interventions: Other: MRI-based techniques; Other: EEG

INTERVENTIONS:
Other: MRI-based techniques — fMRI, DTI
  Other Names: Functional magnetic resonance imaging; Diffusion Tensor Imaging
Other: EEG — ERP
  Other Names: Electroencephaolgraphy; Event-related potential (ERP)

SUMMARY:
Several studies seem to indicate that emotional attention and change-related attention are impaired in ASD. The goal of this study is to identify the relationships between those two types of automatic attention in visual and auditory modalities in subjects with ASD compared to healthy controls and also, over the course of development (children, adults). In order to achieve this goal, the investigators will use complementary techniques (EEG and MRI-based techniques (fMRI, DTI)).

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are characterized by major handicap in social interaction and in daily life adaptation. The orienting response towards potentially relevant events involves automatic attentional mechanisms that would be elicited mainly by two classes of biologically important stimulations: novel stimuli and emotional stimuli. The neural basis of emotional and change-related attention in ASD will be explored by investigating brain reactivity in both visual and auditory modalities, during tasks mixing emotional and non emotional stimuli.

ELIGIBILITY:
Inclusion Criteria:

* No past history of central nervous system disorders
* Written consent
* Affiliated to the National Health Insurance
* Do not participate to another biomedical research
* For ASD group: Children with autism spectrum disorder (DSM-V criteria) and adults with high-functioning autism
* For healthy subjects: No past history of difficulties in early childhood for acquisition of walk, language or reading and no psychiatric disorders

Exclusion Criteria:

* Abnormal corrected vision
* Abnormal audition
* Not stabilized psychoactive treatment or treatment that can modify electrogenesis
* Infectious or metabolic diseases
* Epilepsies
* Impossibility to participate to the whole study
* For subjects participating to the MRI recordings: MRI counter-indications (pace-makers ...), claustrophobia or a positive pregnancy test

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children/ adults with ASD and healthy children/ adults
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05-27 (Actual)

PRIMARY OUTCOMES:
Neural responses to neutral and emotional stimuli | 1 day
  ERP (Event-related potential), fMRI and DTI

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique BONNET-BRILHAULT, MD,PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- University Hospital, Tours, France

REFERENCES:
- [Result] Charpentier J, Kovarski K, Roux S, Houy-Durand E, Saby A, Bonnet-Brilhault F, Latinus M, Gomot M. Brain mechanisms involved in angry prosody change detection in school-age children and adults, revealed by electrophysiology. Cogn Affect Behav Neurosci. 2018 Aug;18(4):748-763. doi: 10.3758/s13415-018-0602-8. PMID 29736682
- [Result] Kovarski K, Latinus M, Charpentier J, Clery H, Roux S, Houy-Durand E, Saby A, Bonnet-Brilhault F, Batty M, Gomot M. Facial Expression Related vMMN: Disentangling Emotional from Neutral Change Detection. Front Hum Neurosci. 2017 Jan 30;11:18. doi: 10.3389/fnhum.2017.00018. eCollection 2017. PMID 28194102
- [Result] Charpentier J, Latinus M, Andersson F, Saby A, Cottier JP, Bonnet-Brilhault F, Houy-Durand E, Gomot M. Brain correlates of emotional prosodic change detection in autism spectrum disorder. Neuroimage Clin. 2020;28:102512. doi: 10.1016/j.nicl.2020.102512. Epub 2020 Nov 27. PMID 33395999
- [Result] Kovarski K, Charpentier J, Roux S, Batty M, Houy-Durand E, Gomot M. Emotional visual mismatch negativity: a joint investigation of social and non-social dimensions in adults with autism. Transl Psychiatry. 2021 Jan 5;11(1):10. doi: 10.1038/s41398-020-01133-5. PMID 33414385
- [Result] Charpentier J, Kovarski K, Houy-Durand E, Malvy J, Saby A, Bonnet-Brilhault F, Latinus M, Gomot M. Emotional prosodic change detection in autism Spectrum disorder: an electrophysiological investigation in children and adults. J Neurodev Disord. 2018 Sep 18;10(1):28. doi: 10.1186/s11689-018-9246-9. PMID 30227832